CLINICAL TRIAL: NCT07314320
Title: A Phase 1, Open-Label, Single-Dose Trial to Evaluate the Mass Balance and Pharmacokinetics of [14C]-OPC-167832 Administered Orally in Healthy Male Subjects
Brief Title: A Study to Detect Radioactivity of [14C]-OPC-167832 in Urine and Feces in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 323-201-00002
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-OPC-167832 (Experimental): Participants receive a single dose of [14C]-OPC-167832, orally, on Day 1.
  Interventions: Drug: [14C]-OPC-167832

INTERVENTIONS:
Drug: [14C]-OPC-167832 — Oral suspension

SUMMARY:
The purpose of this study is to determine the relative amounts of radioactivity excreted in urine and feces following a single oral dose of [14C]-OPC-167832 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 18 to 32 kilograms per square meter (kg/m^2) (inclusive).
2. In good health as determined by:

   1. Medical history
   2. Physical examination
   3. ECG
   4. Serum/urine biochemistry, hematology, and serology tests.
3. Experience regular bowel movements (i.e., at least 1 every day) for 30 days prior to Day -1.
4. Agree to remain exclusively in the research unit for the defined period.
5. Agree to comply with the protocol restrictions and requirements.
6. Ability to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the trial.
7. Male participants and their female partners who commit to remaining abstinent from trial screening through 90 days after the dose of investigational medicinal product (IMP) or utilizing 2 different approved methods of birth control from trial screening through 90 days after the dose of IMP.
8. Commit to refraining from sperm donation from the screening visit through 90 days after the dose of IMP.

Exclusion Criteria:

1. Clinically relevant abnormality in past medical history, or at the screening physical examination, that in the investigator's or sponsor's opinion may place the participant at risk or interfere with outcome variables including distribution, metabolism, and excretion of drug.
2. History of drug and/or alcohol abuse within 2 years prior to screening.
3. History of or current hepatitis or carriers of hepatitis B surface antigen (HBsAg) and/or anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibodies.
4. History of any significant drug allergy or known or suspected hypersensitivity, to any component of the IMP.
5. Participants having taken OPC-167832 within 30 days prior to screening.
6. Participants having 5 half-lives or twice the duration of the biological effect, whichever is longer, of any IMP (inclusive of OPC-167832) within 30 days prior to screening.
7. Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months prior to screening.
8. Any participant who, in the opinion of the investigator, should not participate in the trial.

Note: Other protocol-specified inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Cumulative Amount (Microgram Equivalents) of OPC-167832 Excreted in Urine (Ae,u) | Up to Day 31
Cumulative Amount (Microgram Equivalents) of OPC-167832 Excreted in Feces (Ae,f) | Up to Day 31
Percentage of OPC-167832 Dose Excreted in Urine (%fe,u) | Up to Day 31
Percentage of OPC-167832 Dose Excreted in Feces (%fe,f) | Up to Day 31

SECONDARY OUTCOMES:
Maximum (peak) Concentration (Cmax) of Total Radioactivity in Plasma and Whole Blood | Up to Day 31
Time to Maximum (Peak) Concentration (Tmax) of Total Radioactivity in Plasma and Whole Blood | Up to Day 31
Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Observable Concentration (AUCt) of Total Radioactivity in Plasma and Whole Blood | Up to Day 31
Area Under the Concentration-Time Curve From Time Zero to infinity (AUCinfinity) of Total Radioactivity in Plasma and Whole Blood | Up to Day 31
Terminal-phase Elimination Half-life (t1/2,z) of Total Radioactivity in Plasma and Whole Blood | Up to Day 31
Hemocrit Blood to Plasma Concentration Adjusted Ratio | Up to Day 31
Percentage of Metabolite in Plasma With an AUC > 10% of the AUC of Plasma Radioactivity Based on Radiometric Profiling | Up to Day 31
Cmax of OPC-167832 | Up to Day 31
Tmax of OPC-167832 | Up to Day 31
AUCt of OPC-167832 | Up to Day 31
AUCinfinity of OPC-167832 | Up to Day 31
t1/2,z of OPC-167832 | Up to Day 31
Apparent Clearance (CL/F) of Drug from Plasma Following Extravascular Administration of OPC-167832 | Up to Day 31
Percent Radioactivity Excreted in Urine and Feces as Parent and Identified Metabolites From Profiling data | Up to Day 31
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to Day 31
Number of Participants With Potentially Clinically Relevant Changes in Clinical Laboratory Tests | Up to Day 31
Number of Participants With Potentially Clinically Relevant Changes in Vital Signs | Up to Day 31
Number of Participants With Potentially Clinically Relevant Changes in Physical Examinations | Up to Day 31
Number of Participants With Potentially Clinically Relevant Changes in Electrocardiogram (ECG) Parameters | Up to Day 31

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com/